CLINICAL TRIAL: NCT05615987
Title: Comparison of the Efficacy of 2 Different Botulinum Toxin Injection Techniques in Gastrocnemius Muscle Spasticity in Hemiplegic Patients: A Randomized Double-blind Controlled Study.
Brief Title: Comparison of Botulinum Toxin Injection Techniques in Spasticity
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Konya Beyhekim Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Savaş Karpuz, Medical doctor, Konya Beyhekim Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-01-14
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Spastic Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Botulinum Toxins, Type A; Injections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Classic injection (Active Comparator): 200iu/2ml OnabotulinumtoxinA in total to 2-4 points proximal to the gastrocnemius muscle
  Interventions: Drug: Onabotulinumtoxina for Injection
- İnjection along the length of the muscle (Experimental): A total of 200iu/2ml of onabotulinumtoxinA by spreading along the length of the gastrocnemius muscle
  Interventions: Drug: Onabotulinumtoxina for Injection

INTERVENTIONS:
Drug: Onabotulinumtoxina for Injection — 200iu/2ml in both groups

SUMMARY:
The aim of the study is to compare the effectiveness of the classical (2-4 points to the muscle proximal) application of botulinum toxin in the treatment of spasticity with the application along the length of the gastrecnemius muscle.

The main question it aims to answer Is botulinum toxin more effective in the treatment of spasticity than the classical application applied along the length of the gastrocnemius muscle? Participants will be evaluated for spasticity before and 1 month after injection.

Researchers will compare classical versus application along the length of the muscle to see if there is a reduction in spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with spastic hemiplegia
* Spasticity in the gastrocnemius muscle

Exclusion Criteria:

* Those who have spasticity in other muscles that will affect ankle movements
* Those who use myorelaxant or myospasm-effective drugs
* Those who have been applied botulinum toxin in the last 3 months
* Those who have contractures in the ankle and knee due to orthopedic reasons.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 60 (Estimated)
Dates: Start 2022-12-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2023-10-01 (Estimated)

PRIMARY OUTCOMES:
Spasticity assessment (change between pre-injection and 1-month control) | before injection and 1 month after injection
  Modified ashworth scale
Spasticity assessment (change between pre-injection and 1-month control) | before injection and 1 month after injection
  Tardieu scale
Spasticity assessment (change between pre-injection and 1-month control) | before injection and 1 month after injection
  Joint range of motion measurement
ambulation level (change between pre-injection and 1-month control) | before injection and 1 month after injection
  functional ambulation scale
ambulation velocity (change between pre-injection and 1-month control) | before injection and 1 month after injection
  preferred walking speed

CONTACTS AND LOCATIONS:
Overall Officials: Savaş Karpuz, Principal Investigator — Konya Beyhekim Training and Research Hospital
Locations (1):
- Konya Beyhekim Research and Training Hospital, Konya, Selçuklu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Shared if requested.

REFERENCES:
- [Background] Kim MW, Kim JH, Yang YJ, Ko YJ. Anatomic localization of motor points in gastrocnemius and soleus muscles. Am J Phys Med Rehabil. 2005 Sep;84(9):680-3. doi: 10.1097/01.phm.0000176341.85398.a9. PMID 16141745
- [Background] Prodanov D, Nagelkerke N, Marani E. Spatial clustering analysis in neuroanatomy: applications of different approaches to motor nerve fiber distribution. J Neurosci Methods. 2007 Feb 15;160(1):93-108. doi: 10.1016/j.jneumeth.2006.08.017. Epub 2006 Oct 17. PMID 17049615
- [Background] Shaari CM, Sanders I. Quantifying how location and dose of botulinum toxin injections affect muscle paralysis. Muscle Nerve. 1993 Sep;16(9):964-9. doi: 10.1002/mus.880160913. PMID 8355728
- [Background] Prodanov D, Thil MA, Marani E, Delbeke J, Holsheimer J. Three-dimensional topography of the motor endplates of the rat gastrocnemius muscle. Muscle Nerve. 2005 Sep;32(3):292-302. doi: 10.1002/mus.20378. PMID 15948200
- [Background] Childers MK, Kornegay JN, Aoki R, Otaviani L, Bogan DJ, Petroski G. Evaluating motor end-plate-targeted injections of botulinum toxin type A in a canine model. Muscle Nerve. 1998 May;21(5):653-5. doi: 10.1002/(sici)1097-4598(199805)21:53.0.co;2-w. PMID 9572248
- [Background] Kaymak B, Kara M, Tok F, Ulasli AM, Ozturk GT, Chang KV, Hsiao MY, Hung CY, Yagiz On A, Ozcakar L. Sonographic guide for botulinum toxin injections of the lower limb: EUROMUSCULUS/USPRM spasticity approach. Eur J Phys Rehabil Med. 2018 Jun;54(3):486-498. doi: 10.23736/S1973-9087.17.04667-6. Epub 2017 Apr 4. PMID 28382814
- [Derived] Karpuz S, Yilmaz R, Yilmaz H. Comparison of the Efficacy of 2 Different Botulinum Toxin Injection Techniques in Gastrocnemius Muscle Spasticity in Hemiplegic Patients: A Randomized Double-Blind Controlled Study. Arch Phys Med Rehabil. 2025 Mar;106(3):327-332. doi: 10.1016/j.apmr.2024.09.011. Epub 2024 Sep 27. PMID 39343047